CLINICAL TRIAL: NCT04183543
Title: PEMF Therapy for the Management of Diabetes in Obese Patients (ProMise): A Randomized Controlled Trial
Brief Title: Pemf Therapy for the Management of Diabetes in Obese Patients
Acronym: PROMISE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PROMISE
Record Dates: First submitted 2019-05-24; First posted 2019-12-03 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-06

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: PEMF
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The proposed study is a single-centre, double-blinded randomised controlled trial. Multivariate matching based on gender, age, race and BMI will be carried out before randomisation of one subject in each pair into control or treatment group (matched pairs design). Participants will be excluded if they do not meet all inclusion criteria and/ or meet at least one exclusion criterion. Participants will be randomised 1:1 to either the standard of care/ placebo group (no exposure to fields) or the treatment group (PEMF exposure). The research personnel who are not directly involved in the patient care will prepare a randomisation table. Study research personnel, physicians, dieticians and physiotherapists will be blinded to the randomisation assignment.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulsed Electromagnetic Field Therapy (Experimental): Study participants will receive 20 minutes of PEMFs (10 minutes per leg) on a weekly basis for 16 weeks (Week 1-16). Participants would not be aware of treatment/ sham allocation, as the PEMF device is indistinguishable in operational and non-operational modes. A minimum of 5-day and maximum of 9-day interval between each treatment session shall be followed.
  Interventions: Device: Pulsed Electromagnetic Fields
- Sham Therapy (Sham Comparator): Study participants will receive 20 minutes of placebo treatment (10 minutes per leg) on a weekly basis for 16 weeks (Week 1-16). Participants would not be aware of treatment/ sham allocation, as the PEMF device is indistinguishable in operational and non-operational modes. A minimum of 5-day and maximum of 9-day interval between each treatment session shall be followed.
  Interventions: Device: Sham Therapy

INTERVENTIONS:
Device: Pulsed Electromagnetic Fields — The PEMF device produces pulsed magnetic fields at flux densities up to 1.5 mT peak.
  Arms: Pulsed Electromagnetic Field Therapy
Device: Sham Therapy — Inactive Pulsed Electromagnetic Field therapy
  Arms: Sham Therapy

SUMMARY:
The Investigators previously developed pulsed electromagnetic field stimulation therapy (PEMF) for the metabolic activation of muscle and adipose tissues. In vitro and in vivo preliminary data from rodents demonstrate that PEMF-t induced changes reminiscent of beneficial exercise adaptations, in response to enhanced metabolic fuel utilisation. These exercise mimetic effects were achieved in the absence of exercise and its associated mechanical stresses as the rodents were sedentary. A human pilot study conducted with this platform demonstrated improved muscle function after only 5 weeks.

The PROMISE pilot trial will investigate whether metabolic activation of muscle with a novel, non-invasive technology will further improve metabolic outcomes in overweight/obese patients with early T2DM who are currently given diet and/ or lifestyle interventions.

DETAILED DESCRIPTION:
The modern lifestyle has led to the development and propagation of obesity and type 2 diabetes (T2DM) pandemics. Obesity is associated with increased morbidity and mortality due to its associated diseases such as T2DM; certain cancers; cardiovascular diseases including hypertension, coronary artery disease and stroke; as well as mental disorders. T2DM is currently the main contributor to growing healthcare costs of obesity. One in three Singaporeans is at risk of developing T2DM, and by 2050, this is estimated to cost Singapore about $1.8 billion in medical expenses and productivity lost. With a global population trend towards increased obesity, the prevalence of T2DM will also be increased, thus creating burgeoning health and socioeconomic consequences. An effective interventional strategy against these chronic diseases would not only positively impact human health, but also relieve growing socioeconomic burden.

All guidelines recommend hypocaloric diet and lifestyle interventions (e.g. exercise) to manage T2DM in overweight or obese patients. The goal is to achieve and maintain 5-10%, and 15-20% weight loss in patients with BMI 25-35 kg/m2 and BMI>35 kg/m2, respectively. This goal requires limitation of daily calorie intake to 800-1200 and up to 275 minutes of exercise per week for a moderately obese person. Anti-obesity drugs can also be prescribed for T2DM patients with BMI > 27 kg/m2. When glycaemic control is not achieved, different progressive stages of T2DM are managed by monotherapy, dual therapy and finally triple therapy of Glucose Lowering Drugs (GLDs) without or with insulin program. Invasive bariatric surgeries are also recommended for T2DM patients with BMI >35 kg/m2 (32.5 kg/m2 in Asian populations), as well as lower BMI of 30 - 35 kg/m2 (equivalent to 27.5 - 32.5 kg/m2 in Asian populations) when the metabolic response to regular treatment plans has been poor.

Patient compliance with diet and lifestyle intervention regime can often be challenging, and yet those who faithfully comply may still fail to achieve the necessary weight loss within a limited time-frame. Pharmacotherapy with GLDs also carries some risks for side effects such as hypoglycaemia, weight gain, gastrointestinal problems, infections, bone fracture, pancreatitis, etc. The most effective approach for long term weight loss of >15% and T2DM remission has been bariatric surgery. Hypertension remission rates and metabolic control are also higher with bariatric surgery versus medical treatment. However, surgically treated patients also had significantly higher risk for additional surgical procedures and other complications including abdominal pain, gastroduodenal ulcers, long-term nutrition and micronutrient deficiency, etc. There is a global urgency for patient-friendly yet effective treatment options with minimal side effects for obesity and T2DM.

T2DM remission in bariatric surgery patients has been intricately linked to weight loss. Perhaps most intriguing is the observation that glycaemic control is re-established prior to weight loss and improvement in muscle insulin sensitivity, thus suggesting that there is an earlier mechanistic juncture, potentially amenable to interventional regulation. In the Twin Cycle Hypothesis, fat accumulation in the liver and secondarily in the pancreas, leads to vicious cycles that result in the development of T2DM. Decreasing liver fat content may potentially be the tunable interventional juncture in promoting remission of T2DM in overweight and obese patients. The PROMISE pilot trial will investigate whether metabolic activation of muscle with a novel, non-invasive technology will further improve metabolic outcomes in overweight/obese patients with early T2DM who are currently given diet and/ or lifestyle (DL) interventions.

Better glycaemic control at the early stages of T2DM would

1. improve the management of this progressive disease,
2. reduce reliance on multi-GLDs therapy, and
3. potentially reduce reliance on bariatric surgeries solely for treatment of T2DM.

The Investigators of this study previously developed pulsed electromagnetic field stimulation therapy (PEMF) for the metabolic activation of muscle and adipose tissues. In vitro and in vivo preliminary data from rodents demonstrate that PEMF-t induced changes reminiscent of beneficial exercise adaptations, in response to enhanced metabolic fuel utilisation. These exercise mimetic effects were achieved in the absence of exercise and its associated mechanical stresses as the rodents were sedentary. A human pilot study conducted with this platform demonstrated improved muscle function after only 5 weeks. This study will investigate the use of PEMFs as a non-invasive modality to supplement current clinical standards in enhancing rehabilitation management and improving metabolic outcomes in this clinical base.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Patients who are residing in Singapore for the duration of the study
3. Ability to fulfill follow-up procedure
4. Men and Women aged 30 - 65 years
5. T2DM of duration <10 years (diagnosis based on HbA1c and/or blood glucose)
6. HbA1c ≥ 7% at the last routine clinical check, within the last 12 months if on diet alone
7. HbA1c ≥ 6.5% if on treatment with oral hypoglycemic agent(s)
8. Body Mass Index (BMI) 27.5 - 45 kg/m2
9. Waist circumference < 200 cm (MRI limit)
10. Weight < 200 kg (MRI limit)

Exclusion Criteria:

1. Current insulin use
2. *Current Metformin use
3. Recent HbA1c ≥ 12%
4. Weight loss > 5 kg within the last 6 months
5. Recent eGFR <30 mLs/min/1.73 m2
6. Substance abuse
7. Known cancer
8. Myocardial infarction within the last 6 months
9. Severe heart failure with New York Heart Association (NYHA) grade ≥ 3
10. Current treatment with anti-obesity drug
11. Diagnosed eating disorder or purging
12. Women who are lactating, pregnant or considering pregnancy
13. Patients who have required hospitalisation for depression or are on antipsychotic drugs
14. Patients currently participating in another clinical research trial
15. Patients with contraindications for MR scanning or venipuncture

    * In the event that 80% recruitment cannot be achieved by the end of 2 months, patients on Metformin will be included and prescribed an alternative drug (such as Dipeptidyl peptidase-4 inhibitors (DPP), GLP1 receptor agonist, Sulfonylureas, Alpha glucosidase inhibitor (AGI), or SGLT2 inhibitors) for at least 4 weeks before the start of the trial.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in baseline HbA1c at 17 weeks. | 17 weeks.
  HbA1c will be reported in percentage (%).
Change in baseline fasting blood glucose level at 17 weeks. | 17 weeks.
  Serum glucose will be reported in mmol/L.

SECONDARY OUTCOMES:
Change in baseline serum triglycerides at 17 weeks. | Week 17 (in comparison to baseline measurements).
  Reported in mmol/L.
Change in baseline serum HDL at 17 weeks. | Week 17 (in comparison to baseline measurements).
  HDL is reported in mmol/L.
Change in baseline serum LDL at 17 weeks. | Week 17 (in comparison to baseline measurements).
  LDL is reported in mmol/L.
Change in baseline serum cholesterol at 17 weeks. | 17 weeks.
  Cholesterol is reported in mmol/L.
Change in baseline BMI at 17 weeks. | 17 weeks.
  Weight and height will be combined to report BMI in kg/m^2.
Change in baseline body weight at 17 weeks. | 17 weeks.
  Bodyweight will be measured in kg.
Change in baseline waist-hip ratio at 17 weeks. | 17 weeks.
  Waist and hip circumferences will be measured in cm. Ratio will be calculated as waist measurement divided by hip measurement.
Change in baseline serum C-Peptide at 17 weeks. | 17 weeks.
  C-Peptide will be reported in ug/L
Change in baseline blood pressure at 17 weeks. | 17 weeks.
  BP will be reported in mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Franco-Obregon, Principal Investigator — National University of Singapore; Asim Shabbir, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parate D, Franco-Obregon A, Frohlich J, Beyer C, Abbas AA, Kamarul T, Hui JHP, Yang Z. Enhancement of mesenchymal stem cell chondrogenesis with short-term low intensity pulsed electromagnetic fields. Sci Rep. 2017 Aug 25;7(1):9421. doi: 10.1038/s41598-017-09892-w. PMID 28842627
- [Background] Crocetti S, Beyer C, Schade G, Egli M, Frohlich J, Franco-Obregon A. Low intensity and frequency pulsed electromagnetic fields selectively impair breast cancer cell viability. PLoS One. 2013 Sep 11;8(9):e72944. doi: 10.1371/journal.pone.0072944. eCollection 2013. PMID 24039828
- See also: News article covering MRegen — https://www.straitstimes.com/singapore/health/nus-researchers-create-magnetic-device-to-aid-muscle-recovery